CLINICAL TRIAL: NCT02635048
Title: Efficacy and Safety of Mini-PCNL Versus Standard-PCNL For The Management of 20-40 mm Size Kidney Stones: A Multi-center Randomized Controlled Trial
Brief Title: Mini-PCNL Versus Standard-PCNL For The Management of 20-40 mm Size Kidney Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Baoshan No.2 People's Hospital (Unknown); The Second Affiliated Hospital of Harbin Medical University (Other); First Affiliated Hospital of Fujian Medical University (Other); People's Hospital of Nanhai District, Foshan (Unknown); Yichang Yiling Hospital (Unknown); Suzhou Municipal Hospital (Other); First Affiliated Hospital of Gannan Medical University (Other); General Hospital of Shenyang Military Region (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); The Second Affiliated Hospital of Kunming Medical University (Other); Beijing Chuiyangliu Hospital (Other Government); Fujian Medical University Union Hospital (Other); Shengjing Hospital (Other); 181st hospital of Chinese People's Liberation Army (Other); First Affiliated Hospital of Guangxi Medical University (Other); Jiangmen Central Hospital (Other); China-Japan Union Hospital, Jilin University (Other); The Sixth Affiliated Hospital of Guangzhou Medical University (Other); Jining First People's Hospital (Other)
Responsible Party: Principal Investigator, Guohua Zeng, Vice president, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRER(67)2015
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Kidney Calculi
Keywords: Percutaneous nephrolithotomy; Kidney stones; Efficacy; Safety
MeSH Terms: conditions — Kidney Calculi | interventions — Nephrolithotomy, Percutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Other): Patients in Group 1 undergo mini percutaneous nephrolithotomy
  Interventions: Procedure: Mini Percutaneous Nephrolithotomy
- Group 2 (Other): Patients in Group 2 undergo percutaneous nephrolithotomy
  Interventions: Procedure: Percutaneous Nephrolithotomy

INTERVENTIONS:
Procedure: Mini Percutaneous Nephrolithotomy — patients undergo PNCL with 18Fr nephrostomy tract
  Arms: Group 1
Procedure: Percutaneous Nephrolithotomy — patients undergo PNCL with 24Fr nephrostomy tract
  Arms: Group 2

SUMMARY:
Percutaneous nephrolithotomy (PCNL) has been considered as the first-line choice for the management of >20mm kidney stones. The traditional nephrostomy tract of PNL was dilated to 24-30F, which is referred to as "Standard-PCNL". Standard PNL has an ideal stones free rate (SFR), however, at the cost of severe morbidity. To decrease the disadvantages related to standard PNL, "mini-perc" or "mini-PCNL", 20F or less, was first introduced to pediatric procedure in 1997, and subsequently implemented in adults with the expectation of similar SFR and low morbidity in the past twenty years. Although abundant efforts have been done, whether mini-perc outweigh standard-PNL for the treatment of >20mm calculis in terms of efficiency and safety remains controversial.

To solve this problem, we performed this multicenter, parallel, open-label randomized controlled trial (RCT).

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of mini-PCNL versus standard-PCNL for the management of 20-40 mm size kidney stones.Investigators plan to do a multicenter, parallel, open-label randomized controlled trial (RCT). There are 20 hospitals included in this study, including The First Affiliated Hospital of Guangzhou Medical University, Baoshan No.2 People's Hospital, The second Affiliated Hospital of Harbin Medical University, The First Affiliated Hospital of Fujian Medical University, People's Hospital of Nanhai District, Yichang Yiling Hospital, Suzhou Municipal Hospital, Jining NO.1 People's Hospital, The First Affiliated Hospital of Gannan Medical University, The General Hospital of Shenyang Military, Shanghai General Hospital, Qingyuan People's Hospital, The second Affiliated Hospital of Kunming Medical University, Beijing Chuiyangliu Hospital, Fujian Medical University Union Hospital, ShengJing Hospital of China Medical University, 181st hospital of Chinese People's Liberation Army, The First Affiliated Hospital of Guangxi Medical University, China-Japan Union Hospital, Jilin University, Jiangmen Hospital of Zhongshan University.

Each center performs more than 500 PNL procedures per year. Ethics committee approval was obtained at each site and informed consent was taken from each patient. The primary endpoint was the one-session SFR and the secondary endpoints included intraoperative and postoperative parameters.

This study will be started at January,2016 and ended at November ,2019. The SFR of sPNL and mPNL was assumed to be 83% and 89% respectively, based on the earlier data. -10% was considered as a non-inferiority margin. the type-1 error (α) was set to 0.05 and the power (1-β) to 0.8. Sampling ratio was 1. According to the formulas of 2-sample non-inferiority test comparing two proportions, the minimum sample size for each group was 923 using a power and sample size calculator (HyLown Consulting, Atlanta). Considering the patients lost to follow-up and consent withdrawals, the number was increased to 1000 patients in each group.

Randomization We used SPSS software to generate 2000 random numbers in a table with a ratio of 1:1 ("0" for sPNL and "1" for mPNL). A protocol-blinded coordinator revealed the assignment in sequence to the center once the consent was signed and surgery was scheduled. The number of included patients was not equally distributed among the centers.

Quality control A standard operating procedure (SOP) was made and approved by the principal investigator of each center. Routine monitoring visits to all centers were carried out every month.

Intravenous urography (IVU) and 2 mm non-contrasted CT were done in all patients. CT value was measured with a consistent software in each center. Patients had negative urine culture before treatment. Intravenous single dose of 1st/2nd-generation cephalosporin or ciprofloxacin was administered 30 mins before and after surgery as antibiotic prophylaxis.

All the endoscopic procedures were performed by only one designated experienced surgeon (≥100 procedures per year in both sPNL and mPNL) in each center. All the procedures were performed under general anesthesia and in the prone position. A 5 Fr open-ended ureteral catheter was placed to the renal pelvis through a guide wire. The use of fluoroscopic or/and ultrasonic guidance was determined by the surgeons' preference. An 18-gauge needle was used for puncture. As shown in Fig. 1, the access tract was gradually dilated with fascial introducers (Reborn Medical®) up to 18F (mPNL) or 24F (sPNL). A peel-away sheath was used (Reborn Medical®). The stone was fragmented by pneumatic LithoClast®, or holmium laser with a 550-um laser fiber (Lumenis® and an energy setting of 30-50 W) or ultrasonic lithotripsy (EMS®, only sPNL group). The stone free status was routinely evaluated by fluoroscopy (radiopaque stone) or ultrasound (radio lucent stone). An immediate second-look or another puncture would be performed if needed. A 6 Fr double J stent was inserted for 4 weeks. A 16-18F silastic nephrostomy tube was placed and removed before discharge. Indication for tubeless/total tubeless: absence of major perforation of collecting system, bleeding and/or complete stone clearance.

K.U.B. (kidney-ureter-bladder) plain radiograph and renal ultrasound were used to evaluate the residual stones before discharge. If there was a discrepancy between the presence of residual stones between the KUB and renal ultrasound, a 2 mm non-contrast CT was ordered to better delineate the presence of residual stones and their impact on the clinical management. The status of residual stones was according to the reports assessed by two protocol-blinded radiologists. If the largest residual stone was larger than 6 mm, SWL, RIRS or URL would be recommended before removing double J stent. The one-session SFR (primary outcome) was determined at one month after removing double J stent and defined as either the absence of any residual stone fragments or the presence of clinically insignificant residual stone fragments (CIRFs), without any auxiliary procedures.

The hematocrit drop was measured at 8 am on postoperative day 1. The indications for transfusion was strictly monitored according to the guideline of Chinese Society of Blood Transfusion (hemoglobin less than 70g/l or a progressive decrease in hemoglobin after surgeries). Consideration of angiography and selective angio-embolization for patients with significant macroscopic hematuria in the urine as well as progressive decrease in hemoglobin or unstable hemodynamics. Visual analogue scale (VAS) was used as a pain scale for quantification of postoperative pain at 24h after surgeries.14 VAS was evaluated by two protocol-blinded nurses. Patients with VAS greater than 5 were given nonsteroidal anti-inflammatory drugs. Stone composition was analyzed using uniform instruments (Fourier Transform-Infrared Spectrometry, Thermo®) and method in all participated centers.

Data collection and definitions of parameters The characteristics of patients and clinical outcomes were recorded according to the pre-established case report form (CRF) . Surgical outcomes were predicted preoperatively according to the S·T·O·N·E nephrolithometry. The stone size was the largest diameter of a single stone or the summation of the largest diameters of multiple stones. Operation time was defined as the time from puncture to the placement of the nephrostomy tube or removing the access sheath in cases with tubeless or total tubeless. Septic shock was identified using the clinical criteria of persisting hypotension requiring vasopressor therapy to maintain mean mean artery pressure (MAP) ≥65 mmHg and having a serum lactate level ≥ 2 mmol/L (>18mg/dL) despite adequate fluid resuscitation.

Statistical analysis Statistical analysis was performed using SPSS 20·0. Continuous variables were analyzed using Student's t-test to compare the two means. Categorical variables between groups were analyzed using the chi-squared or Fisher's exact tests. Primary endpoints and some key secondary endpoints were analyzed in both intention-to-treat (ITT) and per-protocol (PP) population. Odds ratio (OR) for sPNL compared with mPNL in categorical variables. Mean difference for sPNL compared with mPNL in continuous variables. P <0·05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients consent for percutaneous renal stone removal
2. Age 18 to 70 years
3. Normal renal function
4. ASA score Ⅰ and Ⅱ
5. Renal stones 20-40mm

Exclusion Criteria:

1. Patients with solitary kidney.
2. Uncorrected coagulopathy and active urinary tract infection (UTI)
3. Morbid obese patients
4. Patients who underwent transplant or urinary diversion.
5. Congenital abnormalities.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1980 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Stone free rate (SFR) | 1 month after removing the pigtail stent
  2mm Non-contrast CT is obtained for all patients at 1 month after removing the pigtail stent to evaluate the final SFR. Stone-free status are defined as either the absence of any residual stone fragments or the presence of clinically insignificant residual stone fragments in the kidney which were defined as ≦ 4mm, asymptomatic, non-obstructive and non-infectious stone particles.

SECONDARY OUTCOMES:
Perioperative complications | intraoperatively or ≤ 1 month postoperatively
  Complication is defined as any adverse event occurred intraoperatively or ≤1 month postoperatively, including intraoperative bleeding, postoperative pain and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Guohua Zeng, PH.D & MD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Department of Urology, Minimally Invasive Surgery Center, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China